CLINICAL TRIAL: NCT03877003
Title: Plasma TMAO and Choline Levels in Individuals With Metabolic Syndrome - Comparison Between Eggs and Choline Supplement Intake
Brief Title: Plasma TMAO and Choline Levels in Individuals With Metabolic Syndrome - Comparison Between Eggs and Choline Supplement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Maria Luz Fernandez, Principal Investigator, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H18-126
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Coronary Artery Disease; Diabetes; Metabolic Syndrome
Keywords: eggs,; choline; metabolic syndrome; TMAO
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Metabolic Syndrome | interventions — Eggs; Dietary Supplements; Choline

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg Intake (Experimental): Consumption of 3 eggs per day for breakfast during 4 weeks
  Interventions: Other: Eggs
- Choline Supplement Intake (Experimental): Consumption of choline supplement 1.5 tablets (approx. 400 mg) with breakfast for 4 weeks
  Interventions: Other: Eggs

INTERVENTIONS:
Other: Eggs — Eggs: Consume 3 eggs per day for 4 weeks Choline supplement: Consume 1.5 pills per day for 4 weeks
  Other Names: Dietary supplement (choline bitartrate)

SUMMARY:
The objective of this study is to determine the effects of consuming either 3 eggs per day and compare it to daily choline supplement (choline bitartrate) for a dose of approximately 400 mg/day on plasma concentrations of high density lipoprotein cholesterol (HDL-c), trimethylamine N oxide (TMAO) and plasma choline. The goal is to determine if choline given as phosphatidyl choline (from eggs) will have a more beneficial effect on plasma choline and microbiota.

DETAILED DESCRIPTION:
Epidemiological data suggests that egg intake does not increase the risk for cardiovascular disease (CVD). In fact eggs are a good source of phosphatidyl choline (PC) and choline has a number of metabolic roles including lipid metabolism, membrane structure, liver health and a neurotransmitter. Recent reports that choline may be metabolized by the intestinal microbiota into TMAO, a compound that may increase the risk for heart disease. It is not clear how much egg contribute to TMAO formation in individuals with metabolic syndrome.

Therefore the objective of this study is to determine the impact of daily intake of 3 eggs versus a choline supplement on plasma TMAO and other biomarkers for CVD risk and also to assess if there are changes in microbiota with these interventions that might lead to the increases of TMAO in plasma.

ELIGIBILITY:
Inclusion Criteria:

* All genders
* 35-70 years
* Metabolic syndrome (based on 3 out of 5 characteristics: waist circumference > 88 cm for women and > 102 cm for men, plasma triglycerides > 150 mg/dL, fasting glucose > 100 mg/dL, blood pressure > 135/85 and HDL < 40 mg/dL for men and < 50 mg/dL for women),
* willing to consume 3 eggs per day for 4 weeks
* willing to consume choline supplement (400 mg/day for 4 weeks)

Exclusion Criteria:

* Self-reported diaberes, cardiovascular disease, history of stroke, liver disease or cancer
* Taking glucose lowering medications
* Taking antibiotics in the previous 1 month
* Triglycerides > 500 mg/dL,
* Cholesterol > 240 mg/dL,
* blood pressure > 145/100 mm of Hg
* Allergic to eggs or to choline

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Plasma choline and TMAO (micromol/L) | 1 year
  They will be measured simultaneously by use of a mass spectrophotometer
Plasma lipids (total cholesterol, HDL cholesterol and triglycerides) in mg/dL | 1 year
  They will be measured simultaneoulsy by use of an automated spectrophotometer

SECONDARY OUTCOMES:
Analysis of microbiota diversity (expressed as concentrations of different microorganisms. | 1 year
  All microorganisms are assayed simultaneously

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Department of Nutritional Sciences, Storrs, Connecticut
  - University of Connecticut, Storrs, Connecticut

IPD SHARING:
Plan to Share IPD: No